CLINICAL TRIAL: NCT04648059
Title: Unmethylated CpG-rich DNA Fragments in TLR-mediated Renal Fibrogenesis of Lupus Nephritis
Brief Title: Epigenetics in Lupus Nephritis
Acronym: Epi_LN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Göttingen (Other)
Collaborators: King's College London (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Peter Korsten, Principal Investigator, University of Göttingen
Other Study IDs: 28/9/17
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: Epigenetics; Methylation; Toll-like receptors; Fibrosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating CpG-rich DNA fragments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lupus nephritis +ve: This group consists of patients with Lupus nephritis
  Interventions: Diagnostic Test: Blood sampling
- Lupus nephritis -ve: This group consist of patients with SLE without Lupus nephritis
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling will be performed to allow analyses of epigenetic markers

SUMMARY:
This is a translational study for the identification of epigenetic changes detectable in sera of patients suffering from Systemic Lupus erythematosus. The aim of the study is to analyze whether circulating DNA fragments are 1) different in patients with or without Lupus nephritis and 2) present and detectable in the circulation before the development of Lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus according to the current classification criteria
* a subgroup requires the presence of Lupus nephritis (no restriction to specific LN histologic subtypes)

Exclusion Criteria:

* patients not able or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of a sample of patients with systemic lupus nephritis (SLE). There will be analyses for the presence of epigenetic markers (methylated CpG-rich DNA fragments) between two groups: 1) patients with SLE with Lupus nephritis (LN) and 2) patients with SLE without LN. In the first phase of the study, a cross-sectional sample of patients will be analyzed. In the second phase of the study, patient samples will be prospectively analyzed for the presence of these markers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Methylated CpG-rich DNA fragments | 12 months
  it will be analyzed whether circulating CpG-rich DNA fragments are present in patients' blood

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No